CLINICAL TRIAL: NCT02441153
Title: T4RC North: Timing of Rectal Cancer Resection After Preoperative Chemoradiotherapy; Does a Longer Wait Improve Outcomes?
Brief Title: Timing of Rectal Cancer Resection After Preoperative Chemoradiotherapy
Acronym: T4RC
Status: Completed | Type: Observational
Sponsor: Health Sciences North Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: T4RC North
Record Dates: First submitted 2015-05-08; First posted 2015-05-12 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2018-02

CONDITIONS: Rectal Neoplasms
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — To maximize the utility of this trial, immunohistochemical staining will be performed on pre-CRT tumor samples to prospectively validate the scoring system proposed by Hur et al. [28] The question being whether or not expression of these biomarkers can predict which patients will experience pCR and disease-free survival.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1(Extended Timing): Surgery will be performed at 10-11 weeks after the completion of chemoradiotherapy.
  Interventions: Other: Extended Timing
- Group 2 (Non-extended timing): Surgery will be performed at 6-7 weeks after completion of chemoradiotherapy.

INTERVENTIONS:
Other: Extended Timing — Surgery will be performed at 10-11 weeks after completion of chemoradiotherapy.
  Groups: Group 1(Extended Timing)

SUMMARY:
This pilot study will take place at Health Sciences North (HSN) in Sudbury. Patients will be identified and screened for inclusion into the study once referred to a general or colorectal surgeon for resection of their rectal cancer. This may occur before or after preoperative chemoradiotherapy (CRT) but randomization will take place after CRT.

DETAILED DESCRIPTION:
The main question of this study is whether or not delaying surgery after preoperative CRT increases disease-free survival. The standard 6-7 week waiting period will be compared to 10-11 weeks, which was the time-frame identified in the Dutch Surgical Colorectal Audit as increasing the likelihood of pCR the most. This trial will also be able to determine if an increased waiting interval increases the rate of sphincter-preservation, local recurrence, and pCR. While similar to the GRECCAR-6 trial, our primary outcome is disease-free survival (a more clinically relevant outcome) and is the first North American clinical trial of this nature.

To maximize the utility of this trial, immunohistochemical staining will be performed on pre-CRT tumor samples to prospectively validate the scoring system proposed by Hur et al. [28] The question being whether or not expression of these biomarkers can predict which patients will experience pCR and disease-free survival.

The pilot will be constructed as a prospective, open-label clinical trial, with patients being randomized to undergo surgery at 6-7 weeks or 10-11 weeks after completion of preoperative CRT. The intention is that once preliminary data is available, other centres in Ontario will be recruited. This will not only help answer our research question, but also create a large, prospective database of rectal cancer patients. The Primary outcome (disease-free survival) will be assessed at 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years)
* T3/4N0M0 or TxN+M0 rectal cancer below or at the peritoneal reflection, confirmed on clinical exam, histology, pelvic MRI, and CT chest/abdo
* Patients who have completed a CRT protocol for the above tumor at HSN
* Informed consent given
* Surgical resection with TME planned

Exclusion Criteria:

* Metastatic disease
* Failure to complete preoperative CRT
* Unable to give free and informed consent
* Unable to comply with the requirements of the study
* Previous malignancy other than nonmelanoma skin cancer, papillary or follicular thyroid cancer
* Inflammatory bowel disease
* Hereditary colorectal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include patients at Health Sciences North who have been referred to a general or colorectal surgeon for resection of their rectal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-12-25 (Actual); Study Completion 2018-01-25 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | 3 years post surgery
  The absence of any local recurrence or metastatic disease discovered on physical exam, endoscopy, or imaging

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Caycedo, MD. M.Sc (c). FRCS. FACS, Principal Investigator — Health Sciences North